CLINICAL TRIAL: NCT02597140
Title: Pilot Study of Effect of Intravenous Lidocaine on Propofol Requirement During Monitored Anesthesia Care in Facial Plastic Surgery
Brief Title: Pilot Study of Effect of Intravenous Lidocaine on Propofol Requirement in Facial Plastic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Responsible Party: Principal Investigator, Chongwha Baek, Professor, Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ChungAng
Record Dates: First submitted 2015-11-03; First posted 2015-11-05 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Anesthesia, Intravenous; Surgery, Plastic
MeSH Terms: interventions — Lidocaine; Saline Solution; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine group (Experimental): Patients will be received an intravenous bolus injection of 1.5 mg/kg lidocaine followed by a continuous lidocaine infusion of 2 mg/kg/hr.
  Interventions: Drug: lidocaine; Drug: propofol
- Control group (Placebo Comparator): Patients will be received an intravenous bolus injection of 1.5 mg/kg normal saline followed by a continuous normal saline infusion of 2 mg/kg/hr.
  Interventions: Drug: normal saline; Drug: propofol

INTERVENTIONS:
Drug: lidocaine — Patients in lidocaine group will be received an intravenous bolus injection of 1.5 mg/kg lidocaine followed by a continuous infusion of 2 mg/kg/hr lidocaine.
  Arms: Lidocaine group
Drug: normal saline — Patients in control group will be received an intravenous bolus injection of 1.5 mg/kg normal saline followed by a continuous infusion of 2 mg/kg/hr normal saline.
  Other Names: 0.9% saline
  Arms: Control group
Drug: propofol — Propofol will be administered using target controlled infusion during monitored anesthesia care to adjust 60 to 80 of bispectral index.
  Other Names: Presofol MCT

SUMMARY:
The purpose of this randomized pilot study is to evaluate the effect of intravenous lidocaine on propofol requirement during BIS (Bispectral index) guided MAC (monitored anesthesia care) in facial plastic surgery.

DETAILED DESCRIPTION:
Several studies reported the usefulness of intravenous lidocaine as a coadjuvant agent during general anesthesia. We thought that there would be an interaction between intravenous lidocaine and hypnotic agent requirement. However, there is no data regarding the effect of systemic lidocaine during MAC. We, thus, would like to perform a randomized, double-blinded pilot study to evaluate the effect of intravenous lidocaine on propofol requirement during BIS guided MAC in facial plastic surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status classification 1 or 2 patients
* aged 20-65 years who were undergoing elective facial plastic surgery under monitored anesthesia care

Exclusion Criteria:

* unwillingness to participate in the study
* adverse reaction to the drugs used in the study
* use of medications that interfere in local anesthetic metabolism
* history of liver disease or kidney failure
* neurological or psychiatric disease
* history of drug or alcohol abuse
* chronic use of benzodiazepine

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
total propofol requirements | during monitored anesthesia care
  Patients' sedation depth will be monitored using a BIS monitor. Propofol will be administered using target controlled infusion (TCI) from targeting 60 to 80 of BIS. At the end of surgery, total propofol requirements will be examined and collected.

SECONDARY OUTCOMES:
postoperative pain | 30 minutes, 2 hours, and 4 hours after surgery
  The outcome assessor will evaluate the degree of postoperative pain using a numeric rating scale (NRS). (0 = no pain, 10 = unimaginable severe pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Ang University Hospital, Seoul, South Korea